CLINICAL TRIAL: NCT06102525
Title: A Phase 1/2a, Open-label, Multicenter, Dose Escalation and Dose Expansion Study Evaluating the Safety, Tolerability, and Efficacy of RZ-001 in Combination With Valganciclovir in Subjects With Glioblastoma
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of RZ-001 With Valganciclovir (VGCV) in Subjects With Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rznomics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RZ-001-201
Record Dates: First submitted 2023-06-23; First posted 2023-10-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1 Cohort 1 (Experimental): RZ-001 Dose 1 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV
- Part 1 Cohort 2 (Experimental): RZ-001 Dose 2 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV
- Part 1 Cohort 3 (Experimental): RZ-001 Dose 3 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV
- Part 1 Cohort 4 (Experimental): RZ-001 Dose 4 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV
- Part 1 Cohort 5 (Experimental): RZ-001 Dose 5 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV
- Part 2 (Experimental): RZ-001 Dose 6 and VGCV
  Interventions: Drug: RZ-001; Combination Product: VGCV

INTERVENTIONS:
Drug: RZ-001 — Recombinant adenovirus harboring the modified ribozyme construct with HSV-tk as a therapeutic transgene
  Other Names: Ad-ECRT-122T
Combination Product: VGCV — VGCV, used in a subject after RZ-001 administration, is a nucleoside analog that is metabolized by HSV-tk and other cellular kinases to form the cytotoxic nucleotide analog ganciclovir triphosphate. An approved oral VGCV will be used in the proposed clinical study of RZ-001.
  Other Names: Valganciclovir

SUMMARY:
This is a Phase 1/2a, open-label study to evaluate the safety, tolerability, immunogenicity, and preliminary clinical activity of RZ-001 administered in combination with VGCV in subjects with hTERT-positive GBM.

DETAILED DESCRIPTION:
The study consists of 2 parts: a dose-escalation part (Part 1) and a dose-expansion part (Part 2).

Part 1 consists of dose escalation exploring MTD/RP2D for intratumoral (IT) injection.

Part 2 will consist of dose expansion exploring clinical activity for the optimal fixed dose based on the results of Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females
* Histologically-confirmed grade 4 astrocytoma, GBM, per The 2021 WHO Classification of CNS Tumors.
* hTERT positive expression confirmed during the screening period
* ECOG score of ≤ 2
* KPS ≥ 60
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Diagnosis of other malignant tumors within 5 years prior to RZ-001 administration.
* Have extracranial metastases of the tumor cells
* Current or history of HIV positive
* Not suitable for inclusion judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | Day 1 to Day 28
Maximum tolerated dose (MTD) or maximum administered dose (MAD) dose(MAD) and select the recommended Phase 2 dose (RP2D) of RZ-001 in combination with VGCV | Day 1 to Day 28
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE | Day 1 to Day 28
  Adverse events (AEs) as characterized by type, number, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE]), timing, seriousness, and relationship to RZ-001
Number of participants with significant laboratory abnormalities as assessed by NCI-CTCAE | Day 1 to Day 28
  Clinically significant laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI-CTCAE), timing, and relationship to RZ-001
Overall survival (OS) | Day 1 to Day 15

SECONDARY OUTCOMES:
Change in concentration of serum vascular endothelial growth factor (VEGF) | Day 1 to Day 28
Change in concentration of serum anti-adenovirus antibody | Day 1 to Day 28
Overall response rate (ORR) | Day 1 to Day 15
Duration of response (DOR) | Day 1 to Day 15
Progression-free survival (PFS) per modified Response Assessment for Neuro-Oncology (mRANO) | Day 1 to Day 15
Overall survival (OS) | Day 1 to Day 15
Neurologic function assessment using the Neurologic Assessment in Neuro-Oncology (NANO) scale ranging from 0 to 3 in each assessment domain | Day 1 to Day 15

OTHER OUTCOMES:
Concentration of adenovirus DNA in Plasma at specified timepoints | Day 1 to Day 28
Change in concentration of serum anti-adenovirus antibody | Day 1 to Day 28
Change in concentration of serum cytokines | Day 1 to Day 28
  Serum cytokines including interleukins 1 (IL-1), IL-6, IL-10, IL-27, interferon gamma (IFN-γ), tumor necrosis factor alpha (TNF-α)
Concentration of biomarker in peripheral blood | Day 1 to Day 28
  Activation of immune cell subsets (including but not limited to cluster of differentiation 3 [CD3], CD4, CD8, B cell, natural killer [NK] cell)
Concentration of biomarker in fresh tumor biopsy tissue | Day 1 to Day 28
  Tumor-related RNA and T cell infiltration and activation

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No